CLINICAL TRIAL: NCT05366933
Title: B-Complex: A Nutraceutical SANS Countermeasure
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Aeronautics and Space Administration (NASA) (U.S. Federal Agency)
Collaborators: Mayo Clinic (Other); Texas A&M University (Other)
Responsible Party: Principal Investigator, Sara R. Zwart, PhD, Deputy Manager for Nutritional Biochemistry, The University of Texas Medical Branch, Galveston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NASA IRB STUDY00000448
Record Dates: First submitted 2022-04-29; First posted 2022-05-09 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Optic Disc Edema; Endothelial Dysfunction
MeSH Terms: conditions — Papilledema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supplemented with B-Complex (Experimental): Subjects will take a vitamin B-complex supplement before, during, and after a 6-12 month spaceflight on the International Space Station
  Interventions: Drug: Vitamin B-Complex Supplement

INTERVENTIONS:
Drug: Vitamin B-Complex Supplement — Vitamin B-Complex Supplement containing: 5-methyltetrahydrofolate, riboflavin 5 phosphate, pyridoxal phosphate, and methylcobalamin

SUMMARY:
In this project, the investigators propose to test effectiveness of a daily nutraceutical supplement containing bioactive B vitamins to mitigate optic disc edema in astronauts. The proposed countermeasure is intended to maximize functioning of the one-carbon metabolic pathway to provide enough substrate and cofactors to overcome any genetic differences that may impact the efficiency of enzyme function. By optimizing the pathway, this will 1) optimize endothelial function by increasing eNOS coupling and nitric oxide synthesis and 2) optimize collagen firmness and elasticity in the sclera and lamina cribrosa, and 3) minimize changes in total retinal thickness during and after flight.

The protocol includes assessments of ocular health and function, along with determinants of vascular endothelial function, advanced glycation end products, and nutritional status and one carbon biochemistry. These additional measures will be critical for the further definition of the causes of optic disc edema in some astronauts after long-duration space flight, and in understanding the effect of the countermeasure. Finally, the supplemented subjects in this study will be compared against total retinal thickness data from previously flown astronauts known to have not taken supplements during their missions.

DETAILED DESCRIPTION:
Fasting (8-h) blood samples (7.5 mL SST and 5 mL EDTA tubes, 12.5 mL total per session) will be collected approximately 180 days and 45 days before flight, on approximate flight day 90, and 30 days before landing, Return to Earth +0-2 days and 30 days after landing.

Blood samples will be analyzed for vitamin status and one-carbon biochemistry, as previously described. One blood sample (collected before flight) will be analyzed for approximately 511 SNPs matching the profile of testing from our ongoing research related to optic disc edema. Serum samples will be analyzed for biochemistry measures evaluating endothelial function, vitamin status, and oxidative damage.

Nutritional status assessment data, including inflight dietary intake and body mass data, completed for routine medical requirements will be requested for data sharing. Inflight medical exercise log data as well as available standard measures data will also be requested for data sharing. Medication use/Med Logs will also be requested for data sharing.

Vascular function VENDYS-II (Endothelix, Inc) will be used to assess reactive hyperaemia through changes in fingertip temperature. The test consists of an automated blood pressure measurement followed by cuff occlusion of the right arm for 2 to 5 min. During this time, the fingertip temperature in the right hand decreases because of the lack of circulation in the fingertip. After the cuff is released, blood flow resumes, causing a temperature rebound in the fingertip in a manner that is proportional to vascular reactivity.

Advanced Glycation End (AGE) Products Skin autofluorescence (SAF) will be analyzed non-invasively using an AGE reader (Diagnoptics Technologies, Groningen, the Netherlands). The AGE reader illuminates a skin surface of approximately 4 cm2, guarded against surrounding light, with an excitation light source with wavelength between 300 and 429 nm. This method is based on the fluorescent properties of certain AGEs accumulated in dermal tissue.

OCT and OCT-A Optical coherence tomography (OCT) and OCT-angiography (OCT-A) scans will be acquired using the Spectralis OCT2 (Heidelberg Engineering) before, during, and after flight. The scan pattern includes 24 B-scans centered in a radial pattern over the optic nerve head, as well as a 3.5 mm circle scan surrounding the optic nerve head for assessment of retinal nerve fiber layer thickness and choroid thickness. For OCT-A, five consecutive volume scans will be obtained in these regions, each containing 216 A-scans. These images will be registered, and the consecutive B-scans will be used to calculate the decorrelation among the images to provide split-spectrum amplitude decorrelation angiography (SSADA) images. This decorrelation between consecutive B-scan images will be used to highlight locations where there is blood flow. The density of the perfused peripapillary vessels within the various layers of the retina will be calculated to create a flow density map.

ELIGIBILITY:
Inclusion Criteria:

• Must be astronauts selected for 6-12 month missions on the International Space Station

Exclusion Criteria:

• Subjects taking B-vitamin supplements

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2032-09-30 (Estimated)

PRIMARY OUTCOMES:
Optic Disc Edema | 6 months
  Measure change in total retinal thickness during and after flight compared to preflight using OCT

SECONDARY OUTCOMES:
Endothelial function | 6 months
  Assess reactive hyperemia through changes in fingertip temperature
Advanced Glycation End Products (AGE) | 6 months
  Skin autofluorescence (SAF) will be analyzed non-invasively using an AGE reader
Serum folate status | 6 months
  Vitamin status assessed from a fasting blood sample
Red Blood Cell folate status | 6 months
  Vitamin status assessed from a fasting blood sample
Vitamin B6 status | 6 months
  Vitamin status assessed from a fasting blood sample
Vitamin B12 status | 6 months
  Vitamin status assessed from a fasting blood sample
Glucose | 6 months
  Serum glucose from a fasting blood sample
Nitric oxide | 6 months
  Serum nitric oxide from a fasting blood sample
tetrahydrobiopterin | 6 months
  Serum biochemistry from a fasting blood sample
Dihydrobiopterin | 6 months
  Serum biochemistry from a fasting blood sample
Oxidized glutathione | 6 months
  Serum biochemistry from a fasting blood sample
Total antioxidant capacity | 6 months
  Serum biochemistry from a fasting blood sample
Advanced glycation end products | 6 months
  Serum biochemistry from a fasting blood sample
Albumin | 6 months
  Serum biochemistry from a fasting blood sample
Glycated albumin | 6 months
  Serum biochemistry from a fasting blood sample
3-nitrotyrosine | 6 months
  Serum biochemistry from a fasting blood sample
Formate | 6 months
  Serum biochemistry from a fasting blood sample
MMP-2 | 6 months
  Serum biochemistry from a fasting blood sample
MMP-9 | 6 months
  Serum biochemistry from a fasting blood sample
TIMP-1 | 6 months
  Serum biochemistry from a fasting blood sample
TIMP-2 | 6 months
  Serum biochemistry from a fasting blood sample
Heparan sulfate | 6 months
  Serum biochemistry from a fasting blood sample
Syndecan-1 | 6 months
  Serum biochemistry from a fasting blood sample
Glypican | 6 months
  Serum biochemistry from a fasting blood sample
Hyaluronan | 6 months
  Serum biochemistry from a fasting blood sample
Total lipid peroxides | 6 months
  Serum biochemistry from a fasting blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Sara R Zwart, PhD, Principal Investigator — UTMB
Locations (1):
- Johnson Space Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zwart SR, Laurie SS, Chen JJ, Macias BR, Lee SMC, Stenger M, Grantham B, Carey K, Young M, Smith SM. Association of Genetics and B Vitamin Status With the Magnitude of Optic Disc Edema During 30-Day Strict Head-Down Tilt Bed Rest. JAMA Ophthalmol. 2019 Oct 1;137(10):1195-1200. doi: 10.1001/jamaophthalmol.2019.3124. PMID 31415055
- [Background] Zwart SR, Gibson CR, Gregory JF, Mader TH, Stover PJ, Zeisel SH, Smith SM. Astronaut ophthalmic syndrome. FASEB J. 2017 Sep;31(9):3746-3756. doi: 10.1096/fj.201700294. Epub 2017 May 25. PMID 28546443
- [Background] Smith SM, Zwart SR. Spaceflight-related ocular changes: the potential role of genetics, and the potential of B vitamins as a countermeasure. Curr Opin Clin Nutr Metab Care. 2018 Nov;21(6):481-488. doi: 10.1097/MCO.0000000000000510. PMID 30169456
- [Background] McGregor HR, Lee JK, Mulder ER, De Dios YE, Beltran NE, Kofman IS, Bloomberg JJ, Mulavara AP, Smith SM, Zwart SR, Seidler RD. Ophthalmic changes in a spaceflight analog are associated with brain functional reorganization. Hum Brain Mapp. 2021 Sep;42(13):4281-4297. doi: 10.1002/hbm.25546. Epub 2021 Jun 9. PMID 34105833
- [Background] Laurie SS, Vizzeri G, Taibbi G, Ferguson CR, Hu X, Lee SMC, Ploutz-Snyder R, Smith SM, Zwart SR, Stenger MB. Effects of short-term mild hypercapnia during head-down tilt on intracranial pressure and ocular structures in healthy human subjects. Physiol Rep. 2017 Jun;5(11):e13302. doi: 10.14814/phy2.13302. PMID 28611153